CLINICAL TRIAL: NCT06871046
Title: An Open-label, Multi-centric Trial to Assess the Safety and Efficacy of an Esflurbiprofen Topical System (EFTS) in the Local Symptomatic and Short-term Treatment of Pain in Contusions.
Brief Title: Phase III Trial to Assess the Safety and Efficacy of TK-254RX in Patients With Contusions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teikoku Seiyaku Co., Ltd. (Industry)
Collaborators: Clinsearch GmbH (Unknown); CRM Biometrics GmbH (Industry); SocraTec R&D GmbH (Other); SocraMetrics GmbH (Industry); HWI pharma services GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TK-254RX-0302; 2024-513064-26-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-10; First posted 2025-03-11 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Contusions
Keywords: Blunt trauma; Soft tissue injuries; sports injuries; NSAIDs; topical patch
MeSH Terms: conditions — Contusions; Wounds, Nonpenetrating; Soft Tissue Injuries; Athletic Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TK-254RX (Experimental): Esflurbiprofen Topical System 165 mg Esflurbiprofen
  Interventions: Drug: Esflurbiprofen Topical System (EFTS)

INTERVENTIONS:
Drug: Esflurbiprofen Topical System (EFTS) — One EFTS is applied to the injured area over 7 days

SUMMARY:
This study is an open-label, multi-centric clinical trial to evaluate the safety and efficacy of TK-254RX in patients with contusions. The primary objective of this study is to assess the safety of TK-254RX. Secondly objective is to evaluate the efficacy of contusions and adhesion of TK-254RX.

ELIGIBILITY:
Inclusion Criteria:

* acute contusion of the upper or lower limbs
* location of injury such that pain-on-movement is elicited on active standardized movement
* enrollment within 6 hours of the injury
* baseline VAS score for POM of injured extremity > 50 mm on a 100 mm VAS
* size of injury, as assessed by Investigator, ≥ 25 cm² and ≤ 120 cm²
* adult male or female patients
* age 18 to 64 years (including)
* having given written informed consent
* satisfactory health as determined by the Investigator based on medical history and physical examination

Exclusion Criteria:

* significant concomitant injury in association with the index soft- tissue injury/contusion; e.g. fracture, nerve injury, ligament disruption, tear of muscle or cartilage, or open wound
* excessively hairy skin at application site, cutting the hair in the injured site prior to patch application will qualify for inclusion
* current skin disorder or shaving hair at application site
* history of excessive sweating/hyperhidrosis inclusive of application site
* intake of NSAIDs or analgesics within 36 hours, opioids within 7 days, or corticosteroids (except inhaled corticosteroids for e.g. topical treatment of bronchial asthma) within 60 days of inclusion in the study
* intake of long-acting NSAIDs or application of topical medication since the injury
* participation in a clinical study within 30 days before inclusion in the study or concomitantly
* participation in this clinical study in another center
* drug or alcohol abuse in the opinion of the Investigator
* pregnant and lactating women
* women of child-bearing potential (defined as all women physiologically capable of becoming pregnant) who are not using an acceptable method of contraception defined as:

  * Surgical sterilization
  * Combined (estrogen and progestogen containing) hormonal contraception, e.g., oral, intravaginal, transdermal and progestogen-only hormonal contraception e.g. oral, injectable, implantable as well as intrauterine device (IUD) and intrauterine hormone-releasing system (IUS) each in combination with male condom to increase safety effect (double barrier method)
  * Total abstinence throughout the study at the discretion of the Investigator.
  * Periodic abstinence is NOT an acceptable method of contraception. An acceptable method of contraception must be maintained throughout the study.
  * A woman who is post-menopausal must have a negative urine pregnancy test at screening but will not need to comply with an acceptable method of contraception. Women are considered post-menopausal and not of child bearing potential if they had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of sterilisation, salpingectomy) or six months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
* known hypersensitivity to Esflurbiprofen, R-flurbiprofen or one of the excipients of the patch
* patients with any ongoing condition that may interfere with the absorption, distribution, metabolism, or excretion of Esflurbiprofen
* history of previous significant injury to the same area within 6 months
* patients with a disease affecting the same area such as synovitis, rheumatoid arthritis, arthrosis, etc.
* patients having an ongoing painful condition associated with blunt injury/contusion
* patients suffering from symptoms of an infectious disease including swelling of any joint of the affected area
* patients who had surgery of the affected area within one year of study entry
* patients with significant diseases (defined as a disease which, in the opinion of the Investigator, may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study; includes patients with a history of gastrointestinal bleeding, significant cardiovascular, liver or renal disease)
* patients with a blood coagulation disorder
* patients who use any impermissible medication
* known allergy to paracetamol and galenic components of the rescue medication

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 221 (Actual)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Recording adverse event and serious adverse event | Day 1 to Day 8
  Characterization of occurence of adverse events or serious adverse events of TK-254RX

SECONDARY OUTCOMES:
100-mm Visual Analogue Scale (VAS) score on pain-on-movement (POM) | Day 1 to Day 8
  VAS score from no pain (0 mm) to worst pain (100 mm) on POM by a patient at each time point
100-mm Visual Analogue Scale (VAS) score on pain-at-rest (PAR) | Day 1 to Day 8
  VAS score from no pain (0 mm) to worst pain (100 mm) on PAR (at least 5 minutes rest) by a patient at each time point
Sum of Pain Intensity Difference (SPID) on pain-on-movement (POM) | Day 1 to Day 8
  Calculating the area under the curve for the difference of each pain intensity score by 100-mm-Visual Analogue Scale (VAS) on movement from the baseline over day 1 to day 8
Sum of Pain Intensity Difference (SPID) on pain-at-rest (PAR) | Day 1 to Day 8
  Calculating the area under the curve for the difference of each pain intensity score by 100-mm-Visual Analogue Scale (VAS) at rest from the baseline over day 1 to day 8
Pain Intensity Difference (PID) on pain-on movement (POM) | Day 1 to Day 8
  Difference of each pain intensity score by VAS on POM from the baseline at each time point
Pain Intensity Difference (PID) on pain-at-rest (PAR) | Day 1 to Day 8
  Difference of each pain intensity score by VAS on PAR form the baseline at each time point
Time to meaningful/optimal reduction | Day 1 to Day 8
  Time to meaningful/optimal reduction of pain defined as first at least 30% (meaningful) and 50% (optimal) reduction from baseline of VAS on POM
Time to complete resolution | Day 1 to Day 8
  * Time to complete resolution of POM VAS value of 0 mm
  * Time to complete resolution of PAR VAS value of 0 mm
Responder rate 1 | Day 3
  Responder rate is defined as the number of patients achieving at least 50% reduction from baseline in the VAS scores for POM at 48 hours
Responder rate 2 | Day 8
  number of patients able to resume training / normal physical activity by 168 hours
Resolution of contusion | Day 8
  The percentage of patients who showed POM=PAR=0 at 168 hours
Global efficacy assessments 1 by investigator | Day 3, Day 4 and Day 8
  The global efficacy assessments are evaluated by the investigator as the response to the following questions: "Considering how this treatment has affected the patient since he/she started in the study, how well is he/she doing?" It is assessed on the following 5-point Likert scale: 0 = very good, 1 = good, 2 = fair, 3 = poor, 4 = very poor.
Global efficacy assessments 2 by investigator | Day 3, Day 4 and Day 8
  The global efficacy assessments are evaluated by the investigator as the response to the following questions: "How would you rate this medication for the treatment of this contution?" It is assessed on the following 5-point Likert scale: 0 = excellent, 1 = very good, 2 = good, 3 = moderate, 4 = poor.
Global efficacy assessments 1 by patients | Day 3, Day 4 and Day 8
  The global efficacy assessments are evaluated by the patients as the response to the following questions: "Considering how this treatment has affected you since you started in the study, how well are you doing?" It is assessed on the following 5-point Likert scale: 0 = very good, 1 = good, 2 = fair, 3 = poor, 4 = very poor.
Global efficacy assessments 2 by patients | Day 3, Day 4 and Day 8
  The global efficacy assessments are evaluated by the patients as the response to the following questions: "How do you rate this medication as a treatment for your contusion?" It is assessed on the following 5-point Likert scale: 0 = excellent, 1 = very good, 2 = good, 3 = fair, 4 = poor.
Characterization of local tolerability | Day 8
  Assessing the local tolerability by using the 8-point dermal response (0: No evidence of irritation, 1: Minimal erythema, barely perceptible, 2: Definite erythema, readily visible, minimal edema or minimal papular response, 3: Erythema and papules, 4: Definite edema, 5: Erythema, edema, and papules, 6: Vesicular eruption, 7: Strong reaction spreading beyond test site) and other effects score (0: No other effect detected, A(0): Slightly glazed appearance, B(1): Markedly glazed appearance, C(2): Glazing with peeling and cracking, F(3): Glazing with fissures, G(3): Film of dried serous exudates covering all or part of the application site, H(3): Small petechial erosions and/or scabs) according to FDA recommendation
Number of use of rescue medication | Day 1 to Day 8
  Number of rescue medication use during clinical study
Patch adhesion assessed by the site staff | Day 2 to Day 5
  Adhesive power of the EFTS will be visually assessed and classified by the site staff in a 5-point-score (0=≥ 90% adhered / 1= ≥75% to <90% adhered / 2=≥50% to <75% adhered / 3=>0% to <50% adhered / 4=completely detached)
Patch adhesion assessed by patient | Day 1 to Day 8
  Adhesive power of the EFTS will be visually assessed and classified by a patient in a 5-point-score (0=≥ 90% adhered / 1= ≥75% to <90% adhered / 2=≥50% to <75% adhered / 3=>0% to <50% adhered / 4=completely detached)

CONTACTS AND LOCATIONS:
Overall Officials: Kenichi Nishiyama, Study Chair — Teikoku Seiyaku Co., Ltd.
Locations (5):
- Germany (5):
  - Medical Practice Ebert, Siemensstr, Bonn
  - Medical Practice Prof. Predel, Siemensstr, Bonn
  - Medical Practice Schaale-Maas, Siemensstr, Bonn
  - Medical Practice Pabst, Sportschule Puch, Fürstenfeldbruck
  - Medical Practice Gastl, Römerstraße, Gilching

IPD SHARING:
Plan to Share IPD: No